CLINICAL TRIAL: NCT05921552
Title: Feasibility of Exercise Prehabilitation Among Older Patients With Hepatobiliary Cancer Planning for Surgery
Brief Title: Senior Adult Hepatobiliary Prehab Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-22153
Record Dates: First submitted 2023-06-16; First posted 2023-06-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Hepatobiliary Cancer; Cholangiocarcinoma; Liver Metastases
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele Health Exercise Prehabilitation (Experimental): Participants will take part in an exercise program in which they will be encouraged to perform approximately 30 minutes of resistance training exercises approximately twice per week until they undergo surgery (Approximately 2-4 weeks). Participants will also be encouraged to perform moderate aerobic exercise such as brisk walking or using stationary aerobic equipment at least 3 times per week. Participants will wear a FitBit fitness watch to monitor aerobic exercise.
  Interventions: Behavioral: Resistance Training; Behavioral: Aerobic Training

INTERVENTIONS:
Behavioral: Resistance Training — Participants will be encouraged to perform approximately 30 minutes of resistance training exercises twice per week, until they undergo surgery. Exercises will be performed using resistance tubes (Bodylastics Inc) and the included accessories (handles and anchor straps) to perform resistance exercises. During Zoom sessions, certified exercise trainers will guide participants to utilize equipment to perform resistance exercises with proper form. Each groups resistance training session will span approximately 1 hour, including a brief warm-up, stretching, and 2 sets of ≥12 repetitions for each of 5 exercises: single arm chest press, single arm row, lateral raise, squat (or chair stand), and resistance tube deadlift.
Behavioral: Aerobic Training — Participants will be encouraged to perform ≥30 minutes of moderate-intensity aerobic exercise on ≥3 days per week. Aerobic exercise intensity will be guided by heart rate zones, with participants exercising at 50-70% of their age-predicted maximum heart rate in bouts of at least 10 minutes at a time. Participants will be encouraged to gradually increase exercise intensity and duration until they are meeting the recommendation

SUMMARY:
The purpose of the study is to evaluate an exercise program for individuals with hepatobiliary cancer planning for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Resectable Hepatocellular carcinoma, Cholangiocarcinoma, or Liver metastasis with Liver resection planned ≥4 weeks
* ECOG 0-2
* Able to sign consent

Exclusion Criteria:

* Does not meet inclusion criteria

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-11-19 (Estimated); Study Completion 2026-11-19 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants that Enroll and Consent - Enrollment Feasibility | Up to 12 Months
  Enrollment will be considered feasible if ≥60% of eligible and approached patients actually consent and enroll
Percentage of Participants that Complete Study Assessments - Retention Feasibility | Up to 3 Months
  Retention will be considered feasible if ≥70% of participants complete study measures
Adherence - Feasibility | Up to 3 Months
  Adherence will be based on participants attending ≥ 70% of tele-RT sessions on average and performing ≥ 70% of prescribed moderate-intensity aerobic exercise per week
Participant Self-Reported Musculoskeletal Injuries - Safety | Up to 3 Months
  The numerator of the safety variable will be the number of musculoskeletal injuries or adverse health events reported as "likely related" or "definitely related" the exercise programming and that caused at least some limitation of daily activity lasting more than 3 days. The denominator for the safety variable will be the number of exercise training sessions attended by the participant.
Exercise Training Safety | Up to 3 Months
  Number of participants that reported any exercise-related musculoskeletal injuries or other adverse health events (e.g.,extreme fatigue, shortness of breath, heat-related illness, cardiovascular events, changes in medication) incurred over the course of the intervention.
Participant Evaluation of Feasibility and Acceptability - Acceptability | Up to 3 Months
  Participants evaluation of feasibility and acceptability will be assessed with a questionnaire, adapted to fit the intervention. The questionnaire includes both Likert Scale and open-ended questions. An item-by-item basis and as average item score, with scores ≥4 ("agree" to "strongly agree") indicating acceptability. Open-ended responses will be analyzed qualitatively to inform intervention improvement.
Objective Physical Functioning and Fitness | At Baseline and Up to 3 Months
  Physical functioning and fitness will be assessed using the 30-second chair stand test,30-second arm curl test, and treadmill 6-minute walk test.
Participant Skeletal Muscle Index (SMI) | At Baseline and Up to 3 Months
  Participants SMI will be measured using Tomovision SliceOMatic software and clinical, computerized tomography (CT) scans
Participants Health-Related Quality of Life | At Baseline and Up to 3 Months
  Participants health-related quality of life will be measured using the 12-item Medical Outcomes Study Short Form Survey
Patient Activation | At Baseline and Up to 3 Months
  Participants patient activation will be measured using the Patient Activation Measure Short Form that is a valid and reliable 13-item scale for measuring patient's self-reported knowledge, skill, and confidence for self-management.
Social Support | At Baseline and Up to 3 Months
  Participants social support will be measured using two scales, the Multidimensional Scale of Perceived Social Support (a valid 12-item measure assessing perceived adequacy of general social support from friends, family, and significant others) and the Social Influence Scale for Exercise (positive influences) (a valid 15-item measure assessing perceived adequacy of exerciserelated social support from friends, family, and experts)
Participant Self Reported Exercise | At Baseline and Up to 3 Months
  Participant self-reported exercise will be measured using a modified Godin Leisure Time Exercise Questionnaire to assess both aerobic and resistance exercise

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Al-Jumayli, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Clinical Trial Search — https://www.moffitt.org/clinicaltrialssearch/?diseasesite=&query=22153&studytype=&medication=&therapy=&pi=&nct=&sortcriteria=